CLINICAL TRIAL: NCT05275972
Title: Descemet Endothelial Thickness Comparison Trials (DETECT I & II)
Brief Title: Descemet Endothelial Thickness Comparison Trial II
Acronym: DETECT II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Oregon Health and Science University (Other); University of California, San Francisco (Other); University of California, Davis (Other); Case Western Reserve University (Other); Dartmouth-Hitchcock Medical Center (Other); University of Pennsylvania (Other); University of Miami (Other); Wills Eye Hospital (Unknown)
Responsible Party: Principal Investigator, Jennifer Rose-Nussbaumer, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20220590-II
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Fuchs; Fuchs Dystrophy; Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — K-115

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DMEK plus topical placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DSO plus topical ripasudil 0.4% (Experimental)
  Interventions: Drug: Ripasudil

INTERVENTIONS:
Drug: Ripasudil — Topical Ripasudil 0.4%
  Arms: DSO plus topical ripasudil 0.4%
Drug: Placebo — Topical Placebo
  Arms: DMEK plus topical placebo

SUMMARY:
Descemet Endothelial Thickness Comparison Trial (DETECT) II is a multi-center, outcome assessor-masked, placebo-controlled clinical trial randomizing 60 patients with Fuchs endothelial dystrophy to DMEK versus Descemet Stripping Only (DSO) with adjunctive Ripasudil.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunctional endothelium from FECD with few guttata extending beyond 4.5 mm
* Peripheral endothelial cell count >1000 cells/mm2 in at least one quadrant
* Good surgical candidate for either procedure as determined by the surgeon
* Willingness to participate
* Age greater than 18 years

Exclusion Criteria:

* Aphakia, anterior chamber IOL or scleral fixated IOL in study eye prior to or anticipated during EK
* Pre-operative central sub-epithelial or stromal scarring that the investigator believes is visually significant and could impact post-operative stromal clarity assessment
* Other primary endothelial dysfunction such as PPMD
* Visually significant optic nerve or macular pathology
* Hypotony (Intraocular pressure <10mmHg)
* Any prior intraocular surgery other than cataract surgery
* >3 clock hours of ANY anterior or posterior synechiae
* >1 quadrant of stromal corneal vascularization
* Inability to comply with post-operative instructions (i.e. unable to position)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Best spectacle-corrected visual acuity (BSCVA) | 12 months
  Best spectacle-corrected visual acuity (BSCVA)

SECONDARY OUTCOMES:
Best spectacle-corrected visual acuity (BSCVA) | 3, 6 and 24 months
  Best spectacle-corrected visual acuity (BSCVA)
Endothelial cell density | 3, 6, and 24 months
  Endothelial cell density

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rose-Nussbaumer, MD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - Stanford University, Palo Alto, California
  - University of California Davis, Sacramento, California
  - University of Miami, Palm Beach Gardens, Florida
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lin CC, Chamberlain W, Benetz BA, Gensheimer W, Li JY, Jeng BH, Clover J, Varnado N, Abdelrahman S, Srinivasan A, Syed ZA, Koo EH, Arnold BF, Lietman TM, Lass J, Rose-Nussbaumer J. Descemet Endothelial Thickness Comparison Trial II (DETECT II): multicentre, outcome assessor-masked, placebo-controlled trial comparing Descemet membrane endothelial keratoplasty (DMEK) to Descemet stripping only (DSO) with adjunctive ripasudil for Fuchs dystrophy. BMJ Open Ophthalmol. 2024 Oct 1;9(1):e001725. doi: 10.1136/bmjophth-2024-001725. PMID 39353677